CLINICAL TRIAL: NCT02423512
Title: The Impact of Anti-TNF Exposure on Vedolizumab Effectiveness: A Biomarker Study.
Brief Title: The Impact of Anti-TNF Exposure on Vedolizumab Effectiveness
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 15-0651; IISR-2015-100947 (Other: Takeda Pharmaceuticals)
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Diseases; Vedolizumab; Ulcerative Colitis; Crohn's Disease; MADCAM1; integrin alpha4beta7
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, mucosal tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anti-TNF Exposure: Inflammatory Bowel Disease (IBD) patients scheduled to start vedolizumab therapy who have been previously exposed to anti-TNF therapy
- anti-TNF Naive: IBD patients scheduled to start vedolizumab therapy who have not been previously exposed to anti-TNF therapy

SUMMARY:
Vedolizumab is a new medication being used for the treatment of Crohn's disease and Ulcerative colitis. It works by blocking specific white blood cells (alpha 4-beta7 lymphocytes) from migrating to areas of inflammation in the gastrointestinal tract. Previous studies have shown that patients who have previous exposure to another type of medication for Crohn's disease and Ulcerative colitis (anti-TNF medications) do not respond to vedolizumab as well as those who have never been exposed. This study will investigate biologic markers in the blood and tissue the help identify possible reasons for this difference.

DETAILED DESCRIPTION:
Patients will be enrolled in the study when they are selected to initiate vedolizumab therapy. Vedolizumab is an intravenous infusion given at increasing intervals. The first infusion of vedolizumab will be considered baseline. Patients may be enrolled at baseline or at colonoscopy prior to the first scheduled infusion of vedolizumab (pre-treatment visit). The standard induction protocol for vedolizumab consists of infusions at week 0 (baseline), week 2, and week 6. Vedolizumab, as per standard-of-care, is then continued at an interval of every 8 weeks following induction therapy. Vedolizumab treatment will be prescribed as per standard practice and will be prescribed regardless of participation in this study. Patients will not receive medication for the sole purpose of this research. Treatment decisions including timing of wash out period between anti-TNf and vedolizumab will be made by the subject's physician and not per the research protocol. There will not be a protocolized washout period for patients previously receiving anti-TNF therapy because treatment will be standard of care and per the directing physician.

Standard of care laboratory tests will be performed by the clinical laboratory at Mount Sinai Hospital. All other measurements will be completed at Prometheus Therapeutics & Diagnostics in San Diego, California or at a Takeda identified lab for vedolizumab concentrations and antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults with a diagnosis of inflammatory bowel disease
* Patients who will be started on vedolizumab therapy as clinically indicated and in discussion with their treating physician will be eligible. Patients will not be started on vedolizumab for the sole purpose of this study

Exclusion Criteria:

-Patients with prior exposure to vedolizumab or natalizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adults with a diagnosis of inflammatory bowel disease who will be started on vedolizumab therapy as clinically indicated and in discussion with their treating physician will be eligible. Patients will not be started on vedolizumab for the sole purpose of this study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
biomarker MAdCAM-1 | baseline and week 14
  change in biomarker MAdCAM-1 at week 14 as compared to baseline

SECONDARY OUTCOMES:
biomarker alpha 4 beta 7 | baseline and week 14
  change in biomarker alpha 4 beta 7 at week 14 as compared to baseline
TNF levels | baseline and week 14
  change in TNF levels at week 14 as compared to baseline
mucosal drug concentration | week 14
  mucosal drug concentration in those undergoing colonoscopy
mucosal drug concentration | week 30
  mucosal drug concentration in those undergoing colonoscopy
vedolizumab drug concentration | week 14
  vedolizumab drug concentration in those patients scheduled for vedolizumab therapy
vedolizumab drug concentration | week 30
  vedolizumab drug concentration in those patients scheduled for vedolizumab therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marla C. Dubinsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Susan and Leonard Feinstein Inflammatory Bowel Disease Center, New York, New York, United States

REFERENCES:
- [Background] Sandborn WJ, Feagan BG, Rutgeerts P, Hanauer S, Colombel JF, Sands BE, Lukas M, Fedorak RN, Lee S, Bressler B, Fox I, Rosario M, Sankoh S, Xu J, Stephens K, Milch C, Parikh A; GEMINI 2 Study Group. Vedolizumab as induction and maintenance therapy for Crohn's disease. N Engl J Med. 2013 Aug 22;369(8):711-21. doi: 10.1056/NEJMoa1215739. PMID 23964933
- [Background] Feagan BG, Rutgeerts P, Sands BE, Hanauer S, Colombel JF, Sandborn WJ, Van Assche G, Axler J, Kim HJ, Danese S, Fox I, Milch C, Sankoh S, Wyant T, Xu J, Parikh A; GEMINI 1 Study Group. Vedolizumab as induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2013 Aug 22;369(8):699-710. doi: 10.1056/NEJMoa1215734. PMID 23964932
- [Background] Sandborn WJ, Colombel JF, Enns R, Feagan BG, Hanauer SB, Lawrance IC, Panaccione R, Sanders M, Schreiber S, Targan S, van Deventer S, Goldblum R, Despain D, Hogge GS, Rutgeerts P; International Efficacy of Natalizumab as Active Crohn's Therapy (ENACT-1) Trial Group; Evaluation of Natalizumab as Continuous Therapy (ENACT-2) Trial Group. Natalizumab induction and maintenance therapy for Crohn's disease. N Engl J Med. 2005 Nov 3;353(18):1912-25. doi: 10.1056/NEJMoa043335. PMID 16267322
- [Background] Sands BE, Feagan BG, Rutgeerts P, Colombel JF, Sandborn WJ, Sy R, D'Haens G, Ben-Horin S, Xu J, Rosario M, Fox I, Parikh A, Milch C, Hanauer S. Effects of vedolizumab induction therapy for patients with Crohn's disease in whom tumor necrosis factor antagonist treatment failed. Gastroenterology. 2014 Sep;147(3):618-627.e3. doi: 10.1053/j.gastro.2014.05.008. Epub 2014 May 21. PMID 24859203
- [Background] Arjis I, De Hertogh G, Machiels K, et al. Mucosal gene expression of cell adhesion molecules, chemokines, and chemokine receptors in patients with inflammatory bowel disease before and after infliximab treatment. American Journal of Gastroenterology. April 2011;106:748-761 Biancheri P, Di Sabatino A, Rovedatti L, et al. Effect of tumor necrosis factor-alpha blockade on mucosal addressin cell-adhesion molecule-1 in Crohn's disease. Inflammatory Bowel Disease. Feb 2013;19(2):259-264.